CLINICAL TRIAL: NCT05574959
Title: Clinical Investigation of the TECNIS® Next-Generation Intraocular Lens, Model DEN00V
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCOL107AHNG
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- investigational Lens Device (Experimental): investigational IOL Model DEN00V
  Interventions: Device: investigational IOL Model DEN00V
- Control Lens Device (Active Comparator): control IOL Model ZCB00/DCB00
  Interventions: Device: control IOL Model ZCB00/DCB00

INTERVENTIONS:
Device: investigational IOL Model DEN00V — Eligible subjects will be randomized in a 1:1 ratio to receive the investigational IOL Model DEN00V in both eyes for the duration of the study.
  Arms: investigational Lens Device
Device: control IOL Model ZCB00/DCB00 — Eligible subjects will be randomized in a 1:1 ratio to receive the control IOL Model ZCB00/DCB00 in both eyes for the duration of the study.
  Arms: Control Lens Device

SUMMARY:
Prospective, multicenter, bilateral, masked (sponsor, subject and evaluator), randomized clinical trial to evaluate the safety and effectiveness of the TECNIS IOL, Model DEN00V in comparison to an aspheric monofocal IOL.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum 22 years of age;
2. Bilateral cataracts for which posterior chamber IOL implantation has been planned;
3. Preoperative best corrected distance visual acuity (BCDVA) of 20/40 Snellen or worse with or without a glare source;
4. Potential for postoperative BCDVA of 20/30 Snellen or better;
5. Corneal astigmatism:

   1. Normal corneal topography;
   2. ≤ 1.0 D of preoperative keratometric astigmatism;
6. Clear intraocular media other than cataract;
7. Availability, ability, willingness and sufficient cognitive awareness to comply with examination procedures;
8. Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries;
9. Ability to understand and respond to a questionnaire in English.

Exclusion Criteria:

1. Requiring an intraocular lens power outside the available range of +14.0 D to +26.0 D;
2. Any clinically significant pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils);
3. Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.);
4. Prior corneal refractive surgery (SMILE, LASIK, LASEK, RK, PRK, etc.);
5. Corneal abnormalities such as stromal, epithelial or endothelial dystrophies that are predicted to cause visual acuity losses to a level worse than 20/30 Snellen during the study;
6. Irregular corneal astigmatism;
7. Inability to achieve keratometric stability for contact lens wearers (as defined in preoperative procedures);
8. History of intraocular surgery, including prophylactic peripheral iridotomies and peripheral laser retinal repairs;
9. Recent ocular trauma that is not resolved/stable or may affect visual outcomes or increase risk to the subject;
10. Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause visual acuity losses to a level worse than 20/30 Snellen during the study;
11. Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration, including pseudoexfoliation, trauma, or posterior capsule defects;
12. Use of systemic or ocular medications that may affect vision;
13. Prior, current, or anticipated use during the 6-month study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) that may, in the opinion of the investigator, confound the outcomes or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery);
14. Poorly controlled diabetes;
15. Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcomes of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.). Note: controlled ocular hypertension without glaucomatous changes (optic nerve cupping and visual field loss) is acceptable;
16. Known ocular disease or pathology that, in the opinion of the investigator:

    1. may affect visual acuity;
    2. may require surgical intervention during the study (macular degeneration, cystoid macular edema, diabetic retinopathy, uncontrolled glaucoma, etc.);
    3. may be expected to require retinal laser treatment or other surgical intervention during the study (macular degeneration, cystoid macular edema, diabetic retinopathy, etc.);
17. Pregnancy, planned pregnancy, presently lactating or another condition associated with hormonal fluctuation that could lead to refractive changes;
18. Concurrent participation or participation within 30 days prior to preoperative visit in any other clinical trial;
19. Desire for monovision correction.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
MONOCULAR PHOTOPIC DCIVA AT 66 CM | at 6-month follow-up
  Mean (logMAR) monocular DCIVA under photopic conditions at 66 cm for first eyes in the investigational vs. control lens groups.
MONOCULAR PHOTOPIC BCDVA AT 4 M | at 6-month follow-up
  Mean (logMAR) monocular BCDVA under photopic conditions at 4 meters for first eyes in the investigational vs. control lens groups.
Secondary Surgical Interventions (SSIs) | at 6-month follow-up
  The rate of Secondary Surgical Interventions (SSIs) related to optical properties of the lens in eyes of subjects in the investigational lens group

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision, Inc. Clinical Trial, Study Director — Johnson & Johnson Surgical Vision, Inc.
Locations (10):
- United States (10):
  - Empire Eye & Laser Center, Bakersfield, California
  - Southern California Eye Physicians and Associates, Long Beach, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Jones Eye Center, Sioux City, Iowa
  - OCLI Vision, Garden City, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Carolina EyeCare Physicians, LLC, Mt. Pleasant, South Carolina
  - Whitsett Vision Group, Houston, Texas
  - Focal Point Vision, San Antonio, Texas
  - Parkhurst NuVision, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu